CLINICAL TRIAL: NCT02089594
Title: Hyperbaric Oxygen Therapy Treatment of Chronic Mild Traumatic Brain Injury (mTBI)/Persistent Post-Concussion Syndrome (PPCS)
Brief Title: Hyperbaric Oxygen Treatment to Treat Mild Traumatic Brain Injury (mTBI)/Persistent Post-Concussion Syndrome (PPCS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul G. Harch, M.D., Clinical Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LSU IRB #7381; W81XWH-10-1-0962 (Other: USAMRMC)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Post-Concussion Syndrome; Traumatic Brain Injury
Keywords: Hyperbaric Oxygen Treatment; Mild Traumatic Brain Injury; Persistent Post-Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Injuries, Traumatic; Brain Concussion | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized prospective controlled
Who Masked: Investigator
Masking Description: Neuropsychological testers and neuropsychologist blinded to treatment group.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric Oxygen Therapy (HBOT) (Experimental): Hyperbaric Oxygen Therapy at 1.5 ATA (atmospheres absolute). The subjects will receive 40 low pressure HBOT's on a once/day, 5d/week eight week schedule.
  Interventions: Drug: Hyperbaric Oxygen
- No Hyperbaric Oxygen Treatment (HBOT) (Experimental): Subjects will receive eight weeks of no hyperbaric treatment while they continue any pre-study maintenance medication and/or pre-study counseling. Subjects will be retested and the control group will be crossed over to receive the identical 40 HBOTs of the HBOT group.
  Interventions: Drug: Hyperbaric Oxygen; Drug: No Hyperbaric Oxygen

INTERVENTIONS:
Drug: Hyperbaric Oxygen — HBOT Group: Pressurization will proceed with 100% oxygen at 1.0 pounds per square inch (psi) per minute, the minimal pressurization rate, to 1.5 ATA (atmospheres absolute) or 7.35 psi and will take approximately 7 minutes. Pressurization will then resume until the final depth of 1.5 ATA is achieved. The patient will remain at depth for approximately 45 minutes and the subject will be informed of the onset of depressurization, which will occur at the same rate as pressurization. Total dive time will be 60 minutes.
  Other Names: Hyperbaric Oxygen Therapy
Drug: No Hyperbaric Oxygen — Subjects will receive their usual care during the equivalent eight-week HBOT treatment period. There will be no hyperbaric chamber experience. At the conclusion of the eight-week control period both control and experimental subjects will be retested and the control group will be crossed over to receive the identical 40 HBOTs of the HBOT group.
  Other Names: Hyperbaric Oxygen Therapy
  Arms: No Hyperbaric Oxygen Treatment (HBOT)

SUMMARY:
Objective/Hypothesis: An eight-week course of forty low-pressure Hyperbaric Oxygen Treatment's (HBOT's) can significantly improve symptoms and cognitive function in subjects with the persistent-post concussion syndrome (PPCS) of mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
This is a randomized prospective controlled single-blind crossover clinical trial of 1.5 ATA (atmospheres absolute) HBOT versus maintenance medication and counseling. One hundred adult subjects (50 at Louisiana State University Health Sciences Center-New Orleans and 50 at Oklahoma State University School of Medicine) with mTBI/PPCS who have been symptomatic continuously for at least six months from one or more mild traumatic brain injuries will be enrolled and randomized to either 40 HBOTs or no treatment. After the 8-week treatment period the no treatment group will be crossed over to receive 40 HBOTs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18-65 years old.
2. One or more mild TBI's due to blunt or blast injury.
3. Meets criteria for PPCS.
4. Ability to complete the NSI.
5. Ability to complete the PCL-M or C.
6. Ability to complete CAPS if needed.
7. Absence of acute cardiac arrest or hemorrhagic shock at time of TBI that would cause a global ischemic insult to the TBI.
8. Ability to complete the Michigan Alcohol Screening Test( MAST) and Drug Abuse Screening Test (DAST).
9. Ability to complete a urine toxicology screen for drugs of abuse.
10. Negative pregnancy test in females. Female subjects will need to have a negative urinalysis result in order to start or continue treatment.
11. Subjects must be legally responsible, speak and understand English fluently, and be able to sign their own consent documents.
12. Otherwise good health.

Exclusion Criteria:

1. Pulmonary disease that precludes HBOT (e.g., bronchospasm unresponsive to medication, bullous emphysema).
2. Unstable medical conditions that are contraindicated in HBOT (e.g. severe congestive heart failure or heart failure requiring hospital emergency evaluation or admission in the previous year).
3. Severe confinement anxiety (e.g., patients who require anesthesia conscious sedation for MRI).
4. Other pre-TBI cerebral neurological diagnoses including stroke, dementia, degenerative diseases, multiple sclerosis, congenital neurological disorder.
5. Participation in another experimental trial with active intervention.
6. High probability of inability to complete the experimental protocol (e.g. terminal condition or inability to complete outcome instruments).
7. Previous HBOT.
8. History of hospitalization for past stroke, non-febrile seizures, or any seizure history other than seizure at the time of TBI.
9. Past or current history of mental retardation.
10. Pre-/post-TBI history of systemic illness with impact on central nervous system (P.I.'s decision).
11. Pre-injury psychiatric disorders for which the patient was on medication at the time of the brain injury responsible for the patient's diagnosis of TBI/PPCS.
12. Any concurrent systemic illness whose symptomatology confounds the diagnosis of PPCS (P.I.'s decision).
13. Active malignancy undergoing treatment.
14. Taking lithium.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Working Memory | One week after final HBOT
Neurobehavioral Symptom Inventory (NSI) | One week after final HBOT

SECONDARY OUTCOMES:
Wechsler Abbreviated Scale of Intelligence II (WASI-II) | 2 months after final HBOT
Wechsler Memory Scale-IV (WMS-IV | 2 months after final HBOT
Rey Auditory Verbal Learning Test (RAVLT) | 2 months after final HBOT
Benton Visual Retention Test with Alternate Forms (Benton VRT) | 2 months after final HBOT
Stroop Color-Word Interference Test | 2 months after final HBOT
Controlled Oral Word Association Test, Letters F, A, and S (COWAT-FAS) | 2 months after final HBOT
Category Fluency Test (Animal) | 2 months after final HBOT
Automated Neuropsychological Assessment Metrics-4 (ANAM-4) | 2 months after final HBOT
Pittsburgh Sleep Quality Index (PSQI) | 2 months after final HBOT
Quality of Life After Brain Injury (QOLIBRI) | 2 months after final HBOT

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Harch, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Louisiana State University Health Sciences Center-New Orleans, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Harch PG, Andrews SR, Rowe CJ, Lischka JR, Townsend MH, Yu Q, Mercante DE. Hyperbaric oxygen therapy for mild traumatic brain injury persistent postconcussion syndrome: a randomized controlled trial. Med Gas Res. 2020 Jan-Mar;10(1):8-20. doi: 10.4103/2045-9912.279978. PMID 32189664